CLINICAL TRIAL: NCT04125589
Title: Understanding The Effects of Acute Stressors and Negative Emotion on Eating Behavior in Binge-Eating Disorder: The Role of Stressor-Induced Changes in Reward and Cognitive Control
Brief Title: Decision Making, Daily Experiences, and Brain Activity in Young Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kristin Nicole Javaras, Assistant Psychologist, Division of Women's Mental Health, McLean Hospital; Assistant Professor of Psychology, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018P001468; K23DK120517 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-10-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Binge-Eating Disorder
Keywords: Binge-Eating Disorder; Decision-Making; Brain Activity
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speaking Activity and Talking Activity (Experimental): Participants will engage in a speaking activity first and a talking activity second.
  Interventions: Behavioral: Speaking Activity; Behavioral: Talking Activity
- Talking Activity and Speaking Activity (Experimental): Participants will engage in a talking activity first and a speaking activity second.
  Interventions: Behavioral: Speaking Activity; Behavioral: Talking Activity

INTERVENTIONS:
Behavioral: Speaking Activity — Participants will engage in a speaking activity where they are given a topic to speak about.
Behavioral: Talking Activity — Participants will engage in a talking activity where they may talk about a topic of their choice.

SUMMARY:
The investigators are doing a study of women with and without binge-eating disorder to learn more about what happens when people engage in everyday decision-making activities. The investigators are interested in learning more about brain activity during everyday decision-making and how everyday decision-making relates to a variety of daily experiences. Examples of everyday decisions include deciding which product to buy, deciding what to eat for a snack, and deciding how to spend free time.

ELIGIBILITY:
INCLUSION CRITERIA:

Inclusion Criteria for All Participants:

* Normal or corrected to normal vision and hearing
* Verbal and written fluency in English
* Right-handed
* Body mass index of 20-35 kg/m^2

Additional Inclusion Criteria for Participants with Binge-Eating Disorder:

• DSM-5 binge-eating disorder

EXCLUSION CRITERIA:

Exclusion Criteria for All Participants:

* Impaired cognition or other neurological/cognitive problems
* Contraindications to MRI (e.g., certain metal implants, claustrophobia)
* Currently/recently/potentially pregnant, seeking to become pregnant in the near future, or breastfeeding
* Serious and/or unstable medical diseases and conditions, and certain other medical diseases and conditions
* Recent low weight
* Certain medications (e.g., insulin)
* Current/recent frequent recreational drug use, or history of frequent recreational drug use in early adolescence
* Extreme dietary limitations (e.g., veganism), pervasive food allergies, or limited exposure to popular snack foods
* Current/recent suicidality
* Current/recent changes in treatment for mental illness
* Study-relevant research experience

Additional Exclusion Criteria for Comparison Participants:

* Personal history of eating disorders or recurrent binge eating
* Personal history of any other mental illness, including serious substance use problems
* First-degree relative with current or past eating or psychotic disorder
* Significant recent change in weight

Additional Exclusion Criteria for Participants with Binge-Eating Disorder:

* Severe mental illness (e.g., psychotic disorder, severe agoraphobia)
* Certain other current/recent mental illness, including severe substance use problems, that would limit study participation or safety
* Recent anorexia nervosa spectrum disorder, avoidant-restrictive food intake disorder, or bulimia nervosa spectrum disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects must identify as female.
Enrollment: 77 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Decision-making behavior (actual decisions) | Up to 1 hour post-intervention
  Decisions (i.e., percent of goal-inconsistent decisions from challenge trials)
Decision-related BOLD activation (reward regions-of-interest) | Up to 1 hour post-intervention
  Percent change in blood oxygen level-dependent (BOLD) signal in response to decision making in regions involved in reward (e.g., nucleus accumbens, insula)
Decision-related BOLD activation (executive function regions-of-interest) | Up to 1 hour post-intervention
  Percent change in blood oxygen level-dependent (BOLD) signal in response to decision making in regions involved in executive function (e.g., dorsolateral prefrontal cortex, inferior frontal gyrus)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin N Javaras, DPhil, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04125589/ICF_000.pdf